CLINICAL TRIAL: NCT06731075
Title: A Double-Blinded, Placebo-controlled, Double Dummy, Multi-center Randomized, Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With Type 2 Diabetes Mellitus With Inadequate Glycemic Control on One to Three Glucose-lowering Agents
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of ORMD-0801 in Subjects With Type 2 Diabetes Mellitus.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oramed, Ltd. (Industry)
Collaborators: InClin, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORA-D-013-3
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Oral Insulin; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ORMD-0801; Insulin

STUDY DESIGN:
Intervention Model Description: In this randomized, double-blind, double dummy, placebo-controlled study, approximately 300 eligible subjects with T2DM and inadequate control on at least one to three glucose-lowering agents will undergo an initial 4-week Screening Period. This will be followed by a 26-week Double-Blind Treatment Period, commencing with a safety Follow-up Visit four weeks after the completion of the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, Contract Reserarch Organization and Medical Laboratories.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ORMD-0801 8 mg once-daily at night - QD (Active Comparator): Double-Dummy; the subject receives both experimental drug and placebo. 1 x 8 mg capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 2 placebo capsules (1 in the morning and 1 at night).
  Interventions: Drug: ORMD-0801 8 mg; Other: Placebo capsule
- ORMD-0801 8 mg twice daily - BID (Active Comparator): Double-Dummy; the subject receives both experimental drug and placebo. 1 x 8 mg capsule each morning approximately 45 minutes (±15 minutes) prior to breakfast and 1 x 8 mg capsule each night prior to bedtime (between 8 PM to 12 Midnight and no sooner than 1 hour after dinner) and 1 placebo capsule at night.
  Interventions: Drug: ORMD-0801 8 mg; Other: Placebo capsule
- ORMD-0801 16 mg once-daily at night - QD (Active Comparator): Double-Dummy; the subject receives both experimental drug and placebo. 2 x 8 mg capsules between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 1 placebo capsule in the morning.
  Interventions: Other: Placebo capsule; Drug: ORMD-0801 16 mg
- Placebo (Placebo Comparator): The subject receives 3 placebo capsules.
  Interventions: Other: Placebo capsule

INTERVENTIONS:
Drug: ORMD-0801 8 mg — 1 x 8 mg capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 2 placebo capsules (1 in the morning and 1 at night).
  Other Names: Oral Insulin
  Arms: ORMD-0801 8 mg once-daily at night - QD; ORMD-0801 8 mg twice daily - BID
Other: Placebo capsule — Placebo capsule
Drug: ORMD-0801 16 mg — 2 x 8 mg capsules between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 1 placebo capsule in the morning.
  Arms: ORMD-0801 16 mg once-daily at night - QD

SUMMARY:
ORA-013-3 is a randomized, controlled study to test the efficacy and safety of an oral capsule of ORMD-0801 at several doses in patients with Type 2 Diabetes Mellitus (T2DM) who have not responded well to other glucose-lowering medications. A total of three hundred subjects will be enrolled in this study and will be required to complete this thirty-four-week clinical trial.

DETAILED DESCRIPTION:
In this randomized, double-blind, double dummy, placebo-controlled study, approximately 300 eligible subjects with T2DM and inadequate control on at least one to three glucose-lowering agents will undergo an initial 4-week Screening Period. This will be followed by a 26-week Double-Blind Treatment Period, commencing with a safety Follow-up Visit four weeks after the completion of the trial. Analysis for the primary and secondary endpoints will be provided for the following subgroups of baseline factors:

1. Sex (Male, Female)
2. Age Group (60 years and younger, over 60 years)
3. Baseline A1C (Less than or equal to 9.0, Greater than 9.0)
4. Race
5. Ethnicity

Screening Period

The Investigator will review the aim of the study, study procedures and potential risks and benefits. These subjects will then sign a written informed consent during the Screening Visit 1 (Screen 1) following which various study procedures will be performed (refer to Table 2). They will be scheduled to return to the clinic 10 days prior to randomization for Screening Visit 2 (Screen 2). At this visit, a CGM sensor will be placed with appropriate instructions by the study team for a 10-day blinded continuous glucose monitoring (CGM) data collection by the site. Subjects will then return to the clinic after 10 days (± 1-day) for removal of the CGM sensor. The subjects will be randomized to one of the four arms of the study treatment.

Treatment Period

After the Screening Period, subjects will be randomized to 26 weeks of Double-Blind Treatment.

In a double-blind, double dummy randomization scheme, subjects will be randomized to one of the following four treatment arms:

1. ORMD-0801 8 mg once-daily at night - QD: 1 x 8 mg capsule between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 2 placebo capsules (1 in the morning and 1 at night).
2. ORMD-0801 8 mg twice daily - BID: 1 x 8 mg capsule each morning approximately 45 minutes (±15 minutes) prior to breakfast and 1 x 8 mg capsule each night prior to bedtime (between 8 PM to 12 Midnight and no sooner than 1 hour after dinner) and 1 placebo capsule at night.
3. ORMD-0801 16 mg once-daily at night - QD: 2 x 8 mg capsules between 8 PM to 12 Midnight and no sooner than 1 hour after dinner and 1 placebo capsule in the morning.
4. Placebo. During the Double-Blind Treatment Period commencing at Week 0 (Visit 1, CGM removal), subjects will return to the clinic at Week 24 - Visit 5 (10 days prior to Week 26 for CGM application) and Week 26 - Visit 6 (CGM removal and end of Double-Blind Treatment Period visit).

The visit requiring CGM application will occur 10 days prior to the CGM removal visit within ± 1-day window.

Safety Follow-up/End of Study All subjects completing the trial will return to the clinic in 4 weeks ± 3 days for a safety Follow-up Visit. Study procedures and assessments will be performed.

Subjects withdrawing prematurely from the trial will have the early termination (ET) visit procedures completed. All patients will continue to be followed in accordance with ITT principles to avoid lost to follow-up and missing data.

Throughout the course of the study, subjects will measure and record fasting blood glucose levels at least 2-3 times a week [self-monitored blood glucose (SMBG)] or when they experience any symptoms of hypoglycemia using a glucose meter. Subjects will be provided a paper diary at each clinic visit and trained to record information related to fasting blood glucose and description of hypoglycemic events: time and date of occurrence; symptoms experienced, if any; treatment given, if any; and specific circumstances. Subjects will be required to bring the paper diary at each clinic visit where data will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 50 years.
* Established diagnosis of T2DM for at least 6 months prior to Screening AND an A1C ≥ 7.2% but ≤ 10.0% at Screening.
* On a stable dose of at least one and up to three of the following glucose-lowering agents: Metformin, sulfonylurea, DPP-4 inhibitor, SGLT-2 inhibitor, thiazolidinedione, insulin secretagogue, oral or injected GLP-1 receptor agonists, glucosidase inhibitor, or pramlintide (injected insulin is excluded) for a minimum of 3 months prior to Screening.
* Body mass index (BMI) of ≤ 28 kg/m2 at Screening and stable weight, with no more than 5 kg gain or loss in the 3 months prior to Screening.
* Renal function - eGFR ≥ 30 ml/min.
* Females of childbearing potential must:
* - a. Have a negative serum pregnancy test result at Screening.
* - b. Agree to avoid becoming pregnant while receiving IP for at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP.
* - c. Agree to use an acceptable method of contraception at least 30 days prior to IP administration, during the entire study, and for 30 days following their last dose of IP. Acceptable methods of contraception are hormonal contraception (contraceptive pill or injection) PLUS an additional barrier method of contraception such as a diaphragm, condom, sponge, or spermicide.
* - d. In the absence of hormonal contraception, double-barrier methods must be used which include a combination of any two of the following: diaphragm, condom, copper intrauterine device, sponge, or spermicide, and must be used for at least 30 days prior to administration of IP, during the entire study, and for 30 days following their last dose of IP.
* - e. Abstinence (relative to heterosexual activity) can be used as the sole method of contraception if it is consistently employed as the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ERCs/IRBs. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.
* - f. Females who are not of childbearing potential are defined as:
* - - - - - i. Postmenopausal (defined as at least 12 months with no menses in women ≥ 45 years of age); OR
* - - - - - ii. Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal ligation/occlusion at least 6 weeks prior to screening; OR
* - - - - - iii. Have a congenital or acquired condition that prevents childbearing.

Exclusion Criteria:

* Type 1 diabetes by history.
* Diabetes attributable to other secondary causes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant).
* Treatment involving injected insulin within 3 months prior to Visit 1.
* A history of > 2 episodes of severe hypoglycemia within 6 months prior to Screening.
* A history of hypoglycemic unawareness.
* A history of unstable angina or myocardial infarction within 6 months prior to Screening, New York Heart Association (NYHA) Grade 3 or 4 congestive heart failure (CHF), valvular heart disease, ventricular cardiac arrhythmia requiring treatment, pulmonary hypertension, cardiac surgery, coronary angioplasty, stroke, or transient ischemic attack (TIA) within 6 months prior to Screening.
* A history of uncontrolled or untreated severe hypertension defined as systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg. A single repeat measurement will be permitted
* Renal dysfunction: eGFR < 30 mL/min.
* A history of or active proliferative retinopathy requiring treatment.
* Psychiatric disorders that, per Investigator judgment, may have impact on the safety of the subject or interfere with subject's participation or compliance in the study.
* Laboratory abnormalities at Screening including:
* - - a. Abnormal serum thyrotropin (TSH) levels below the lower limit of normal or >1.5X the upper limit of normal; a single repeat test is allowable.
* - - b. Elevated liver enzymes (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP)) > 3X the upper limit of normal; a single repeat test is allowable.
* - - c. Very elevated fasting triglyceride levels (> 600 mg/dL); a single repeat test is allowable.
* - - d. Any relevant abnormality that would interfere with the efficacy or the safety assessments during study treatment administration.
* Positive history of active liver disease (other than non-alcoholic hepatic steatosis), primary biliary cirrhosis, or active symptomatic gallbladder disease.
* Positive results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus ribonucleic acid (RNA).
* Patient has active or history of neoplastic disease (except for adequately treated non-invasive basal cell and/or squamous cell carcinoma or carcinoma in situ of the cervix) within the past 5 years prior to baseline.
* Use of the following medications:
* - - -a. History of use of any injectable insulin (greater than 7 days) within 6 months prior to Screening.
* - - -b. Administration of thyroid preparations or thyroxine (except in subjects on stable replacement therapy) within 6 weeks prior to Screening.
* - - - c. Use of oral, intravenous, or intramuscular steroids for one month prior to enrollment. Intra-articular and/or topical corticosteroids are not considered systemic.
* - - - d. Concurrent use of medications known to modify glucose metabolism or to decrease the ability to recover from hypoglycemia such as oral, parenteral, and immunosuppressive or immunomodulating agents. Inhaled nasal steroids are permissible.
* Known allergy to soy.
* Involvement in a weight loss program and is not in the maintenance phase, or subject has started weight loss medication (e.g., orlistat or liraglutide) within 3 months prior to Screening.
* Prior bariatric surgery.
* Subject is pregnant or breast-feeding.
* Subject is a user of recreational or illicit drugs or has had a recent history (within 1 year of Screening) of drug or alcohol abuse or dependence. (Note: Alcohol abuse includes heavy alcohol intake as defined by > 3 drinks per day or > 14 drinks per week or binge drinking) at Screening. Occasional intermittent use of cannabinoid products will be allowed provided that no cannabinoid products have been used during the 1 week prior to each visit.
* Weight loss preparations either approved and marketed or used in OTC preparations except for GLP-1 used in the treatment of underlying diabetes.
* Any condition or other factor (at the Investigator's discretion) that is deemed unsuitable for subject enrollment into the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in A1C at 26 weeks | Visit 1 (baseline) and Visit 6 (week 26)
  Change from baseline (Visit 1) in A1C at 26 weeks (Visit 6).

SECONDARY OUTCOMES:
Incidence of A1C < 7% at 26 weeks (Visit 6). | Week 26
  Number of subjects that have a value of A1C less than 7%
Change from baseline in fasting plasma glucose at week 26 | Baseline (Visit 1) to Week 26 (Visit 6)
  Change from baseline in fasting plasma glucose (FPG) at week 26
Safety Assessment by number of adverse events. | Visit 1 (baseline) through Visit 6 (week 26)
  Safety assessed by number of adverse events including adverse events of special interest such as hypoglycemia.

OTHER OUTCOMES:
Changes from baseline over time for A1C | Measurements between Visit 1 (baseline) and Visit 6 (week 26)
  Changes from baseline over time for A1C and during the Double-Blind Treatment Period.
Changes from baseline over time for FPG | Measurements between Visit 1 (baseline) and Visit 6 (week 26)
  Changes from baseline over time for FPG during the Double-Blind Treatment Period.
Change of Mean Sensor Glucose, | Baseline (Visit 1) to Week 26 (Visit 6)
  Change in CGM Mean Sensor Glucose from baseline to week 26.
Time in Range (TIR) of Sensor Glucose < 54 mg/dL | Baseline (Visit 1) to Week 26 (Visit 6)
  Time in Range duration of CGM Sensor Glucose when Sensor Glucose falls in the range of < 54 mg/dL
Time in Range (TIR) of Sensor Glucose 54-69 mg/dL | Baseline (Visit 1) to Week 26 (Visit 6)
  Time in Range duration of CGM Sensor Glucose when Sensor Glucose falls in the range of 54-69 mg/dL
Time in Range (TIR) of Sensor Glucose 70-180 mg/dL | Baseline (Visit 1) to Week 26 (Visit 6)
  Time in Range duration of CGM Sensor Glucose when Sensor Glucose falls in the range of 70-180 mg/dL
Time in Range (TIR) of Sensor Glucose 180-250 mg/dL | Baseline (Visit 1) to Week 26 (Visit 6)
  Time in Range duration of CGM Sensor Glucose when Sensor Glucose falls in the range of 180-250 mg/dL
Time in Range (TIR) of Sensor Glucose >250 mg/dL | Baseline (Visit 1) to Week 26 (Visit 6)
  Time in Range duration of CGM Sensor Glucose when Sensor Glucose falls in the range of >250 mg/dL
Incidence of A1C < 8% at 26 weeks | 26 Weeks (Visit 6)
  Incidence of A1C < 8% at 26 weeks (Visit 6).
Incidence rate of subjects requiring glycemic rescue therapy and the time to rescue. | Baseline (Visit1) through Week 26 (Visit 6)
  Incidence rate of subjects requiring glycemic rescue therapy and the time to rescue during the Double-Blind Treatment Period.
Change in weight from baseline | Baseline (Visit 1) and Week 26 (Visit 6)
  Change in weight from baseline during the Double-Blind Treatment Period.
Changes from baseline over time for C-peptide | Baseline (Visit 1) through Week 26 (Visit 6)
  Changes from baseline over time for C-peptide during the Double-Blind Treatment Period.
Changes from baseline over time in fasting insulin | Baseline (Visit 1) through Week 26 (Visit 6)
  Changes from baseline over time in fasting insulin during the Double-Blind Treatment Period.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kidron, Ph.D., Study Director — Oramed, Ltd.
Locations (1):
- Velocity Clinical Research Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized IPD will be shared.

REFERENCES:
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Nathan DM, Buse JB, Davidson MB, Heine RJ, Holman RR, Sherwin R, Zinman B. Management of hyperglycemia in type 2 diabetes: A consensus algorithm for the initiation and adjustment of therapy: a consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2006 Aug;29(8):1963-72. doi: 10.2337/dc06-9912. No abstract available. PMID 16873813
- [Background] Li X, Yang S, Cao C, Yan X, Zheng L, Zheng L, Da J, Tang X, Ji L, Yang X, Zhou Z. Validation of the Swedish Diabetes Re-Grouping Scheme in Adult-Onset Diabetes in China. J Clin Endocrinol Metab. 2020 Oct 1;105(10):dgaa524. doi: 10.1210/clinem/dgaa524. PMID 32808015
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 3. Prevention or Delay of Type 2 Diabetes and Associated Comorbidities: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S41-S48. doi: 10.2337/dc23-S003. PMID 36507633
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Cleary PA, Orchard TJ, Genuth S, Wong ND, Detrano R, Backlund JY, Zinman B, Jacobson A, Sun W, Lachin JM, Nathan DM; DCCT/EDIC Research Group. The effect of intensive glycemic treatment on coronary artery calcification in type 1 diabetic participants of the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study. Diabetes. 2006 Dec;55(12):3556-65. doi: 10.2337/db06-0653. PMID 17130504
- [Background] Mansour Aly D, Dwivedi OP, Prasad RB, Karajamaki A, Hjort R, Thangam M, Akerlund M, Mahajan A, Udler MS, Florez JC, McCarthy MI; Regeneron Genetics Center; Brosnan J, Melander O, Carlsson S, Hansson O, Tuomi T, Groop L, Ahlqvist E. Genome-wide association analyses highlight etiological differences underlying newly defined subtypes of diabetes. Nat Genet. 2021 Nov;53(11):1534-1542. doi: 10.1038/s41588-021-00948-2. Epub 2021 Nov 4. PMID 34737425